CLINICAL TRIAL: NCT01106170
Title: A Double-Blind, Placebo-Controlled, Crossover Evaluation of a Grape Seed Extract and Quercetin Supplement (Provex CV) to Reduce Markers of Inflammatory Cytokines and Blood Pressure in Subjects With Metabolic Syndrome
Brief Title: Efficacy of Provex CV Supplement to Reduce Inflammation Cytokines and Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 31886 Melaluca-ProvexCV
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Participants will consume 330 mg of Provex CV supplement, by mouth, per day, for 4 weeks followed by 4 weeks of 330 mg of placebo (cornstarch)
  Interventions: Drug: Provex CV; Other: placebo
- Arm 2 (Experimental): Participants will consume 330 mg placebo (cornstarch), by mouth, per day for 4 weeks followed by 4 weeks of 330 mg of ProvexCV for 4 weeks.
  Interventions: Drug: Provex CV; Other: placebo

INTERVENTIONS:
Drug: Provex CV — dietary supplement, 2 capsules per day by mouth
Other: placebo — corn starch, 2 capsules per day by mouth

SUMMARY:
The purpose of this study is to determine if a supplement called Provex CV can reduce blood pressure and other risk factors for heart disease. Heart disease is the leading cause of death in this country and it is important to identify dietary factors, including supplements, that can reduce heart disease risk factors. The supplement to be tested in this study is made of a combination of natural compounds found in plants such as grapeseed extract, green tea, and quercetin. Each compound individually has been shown to improve blood pressure or reduce inflammation. We hypothesize that Provex CV will reduce blood pressure and levels of inflammatory cytokines hypertensive patients with symptoms of metabolic syndrome. This investigational trial of Provex CV has been approved by the United States Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Males (18 - 65) and postmenopausal females (up to age 65) with metabolic syndrome who have stage 1 hypertension.
* Since all subjects will have Stage 1 hypertension, they must also meet at least 2 of the following criteria of metabolic syndrome to qualify for the study; waist circumference of >35 inches for women or >40 inches in men, fasting plasma triglycerides of >150 mg/dl, fasting glucose of >100 mg/dl, HDL of <40 in men. Pre-hypertension or greater (130 + mm Hg systolic/80+mm Hg diastolic) is defined by the 7th Report for the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure.

Exclusion Criteria:

* Subjects who are allergic to tea or grapes (on which the supplement is based).
* Participants who have blood pressure less than 130 mmHg / 80 mmHg,
* have a history of a prior cardiovascular event, diabetes, pregnancy, liver disease, renal insufficiency, any chronic disease that might interfere with study participation,
* BMI above 40 kg/m2,
* consumption of >12 alcoholic drinks weekly,
* unwillingness to stop current supplement intake or use of calcium/ magnesium antacids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 weeks after supplement or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thunder Jalili, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Biesinger S, Michaels HA, Quadros AS, Qian Y, Rabovsky AB, Badger RS, Jalili T. A combination of isolated phytochemicals and botanical extracts lowers diastolic blood pressure in a randomized controlled trial of hypertensive subjects. Eur J Clin Nutr. 2016 Jan;70(1):10-6. doi: 10.1038/ejcn.2015.88. Epub 2015 Jun 10. PMID 26059745